CLINICAL TRIAL: NCT05281835
Title: Follow-up of Elderly Subjects With Falls Recruited in the Geriatric Departments of Several French Hospitals
Acronym: PREMOB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_90; 2021-A00582-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Falls in the Elderly
Keywords: Elderly; Fallers; Falls; Risk factors; Cohort; National Health Data System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Falls are the leading cause of accidental death among the elderly, with nearly 8,000 deaths per year in France, including more than 950 deaths on average per year in the Northwest interregion between 2006 and 2013. The incidence of falls increases with age. Falls are often the consequence of multiple factors: extrinsic and intrinsic. The WHO classifies these risk factors into 4 groups: environmental, socio-economic, behavioral and biological.

The best way to act to reduce falls is to identify the risk and severity factors (risk of fracture, risk of loss of autonomy, risk of death) in order to correct those that are modifiable.

On a national scale, the prevention of falls has been considered for many years as a major issue in health prevention [INPES 2005]. The management of elderly patients who fall has been the subject of recommendations for good practice by the French National Authority for Health (HAS) in 2009. These recommendations include the need to look for signs of geriatric severity of falls.

The SNDS National System of healthcare data brings together and links the main national health databases in France. Linking data from the PMSI (Programme de Médicalisation des Systèmes d'Information) and the National Inter-regime Information System of the French National Health Insurance with data from death certificates via the SNDS opens up unique perspectives for improving the quality of follow-up of these patients. Crossing data from the Fall assessment clinic (clinical data) and SNDS data will allow data completeness and will improve our knowledge of the care consumption of elderly fallers. In particular, we wish to determine the risk factors for unplanned hospitalizations of patients with falls.

This project aims to set up a common multicenter cohort of patients assessed during the day hospital for multidisciplinary fall assessment in 12 geriatric services: the university hospitals of Lille, Amiens-Picardie, Rouen, Caen, Tours, Strasbourg, Angers, Dijon, the GHICL and the hospitals of St Quentin, Valenciennes and Beauvais Data collection is currently being harmonized in all participating clinical departments. The databases of the SNDS and that of the fall day hospital assessment will be crossed. This will allow us to improve our knowledge of the follow-up of elderly fallers, the impact of risk factors (clinical, psychosocial, organizational, etc.) and their interactions, the effectiveness of specific management on the occurrence of falls, serious falls as well as the use of care. 1,000 elderly patients admitted in 12 French geriatric departements for a fall assessment will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 65 years of age or older
2. Patients admitted at a day hospital for multidisciplinary falls assessment in one of the 12 geriatric department participating in the study
3. Patient or, if applicable, his or her trusted person or guardian, having given his or her oral non-opposition
4. Patient affiliated to a social health insurance scheme (beneficiaries or beneficiaries' dependents)

Exclusion Criteria:

1. Expressed objection to the collection of data by the subject, his or her guardian, curator, trusted person or family member.
2. Admission at the day hospital for multidisciplinary falls assessment is not indicated (despite the referral of the patient and the realization of the initial consultation).
3. Refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients admitted at a day hospital for multidisciplinary falls assessment in one of the 12 french geriatric department participating in the study
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the first unplanned hospitalization within 1 year after the day hospital for multidisciplinary falls assessment | 1 year of follow up

SECONDARY OUTCOMES:
Time between initial consultation (HDJ fall) and 1st unscheduled hospitalization occurring within 12 months of follow-up (dependent variable) and potential predictive factors | within 12 months
  Time between initial consultation (HDJ fall) and 1st unscheduled hospitalization occurring within 12 months of follow-up (dependent variable) and potential predictive factors (independent variables): behavioral, environmental, medical-biological and socioeconomic factors.
Number of unplanned hospitalizations during the 12 months of follow-up or until the patient's death (expressed as number of hospitalizations per 100 patient years). | within 12 months
Time from initial consultation (HDJ fall) to occurrence of death within 12 months of follow-up. | within 12 months
Time between the initial consultation (HDJ fall) and the first hospitalization for fracture during the 12 months of follow-up. | within 12 months
Time from initial consultation (HDJ fall) to occurrence of 1st unplanned hospitalization or death within 12 months of follow-up. | within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François Puissieux, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Usld Les Bateliers Chr Lille - Lille, Lille, France